CLINICAL TRIAL: NCT04167254
Title: Feasibility of Implementing Sit Down and Play in Routine Visits in India
Brief Title: Sit Down and Play India
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Reshma Shah, MD, Assistant Professor of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-0337_4
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Development, Child

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sit Down and Play (Experimental)
  Interventions: Behavioral: Sit Down and Play
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Sit Down and Play — Brief health care-based program that aims to promote key parenting behaviors that promote early childhood development
  Arms: Sit Down and Play

SUMMARY:
To gather data essential to evaluate the acceptability and feasibility of a brief, health care-based program delivered in routine healthcare visits in low and low-middle income countries to promote positive parenting behaviors with the aim to support early child development.

ELIGIBILITY:
Inclusion Criteria:

Parents/legal guardians will be eligible if they:

* Are over the age of 18 years
* Have a child between 6 and 10 weeks
* Are presenting to Deshnur and Murgod Primary Health Centers in Karnataka, India for a heatlh visit and
* Self-identify as the "primary caregiver.

Exclusion Criteria:

Parents/legal guardians will be ineligible if they:

* Are less than the age of 18 years
* Have a child who is not between 6 and 10 weeks or
* Have a child who is sick at the time of visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Parenting Behaviors that Promote Early Childhood developme | 1 month after second immunization visit
  Key items from the UNICEF Multiple Indicator Cluster Surveys Early Childhood Development Module

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Shah, Principal Investigator — University of Illinois at Chicago
Locations (2):
- University of Illinois at Chicago, Chicago, Illinois, United States
- Deshnur Primary Health Center, Deshnur, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah R, Herekar V, Metgud D, Kim H, Atkins M, Dhaded S. Implementing an early childhood development intervention with routine immunization visits in India: a feasibility trial. Eur J Pediatr. 2022 Jul;181(7):2799-2808. doi: 10.1007/s00431-022-04485-w. Epub 2022 May 5. PMID 35508559